CLINICAL TRIAL: NCT00094939
Title: Predictors of Cognitive Decline in Normal Aging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Other Study IDs: IA0056; R01AG012101 (NIH)
Record Dates: First submitted 2004-10-28; First posted 2004-10-29 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-09

CONDITIONS: Alzheimer Disease; Dementia
Keywords: mild cognitive impairment; Alzheimer disease; magnetic resonance imaging; CSF tau protein; Hippocampus
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The goal of this project is to develop an early diagnostic test for Alzheimer's disease (AD) by monitoring loss of neurons and brain size reductions over a period of five years.

DETAILED DESCRIPTION:
Studies of normal aging and mild cognitive impairment (MCI) show that loss of neurons and reduction in size of the hippocampal part of the brain predict a person's conversion from MCI to Alzheimer's disease (AD). Increases in tangle-related abnormal tau proteins, specifically P-tau231, also appear to be related.

This study will collect neuropsychological data, magnetic resonance imaging (MRI), and cerebrospinal fluid (CSF) from volunteer participants to measure the relationship between changes in brain volume, CSF levels, and memory performance.

From the data researchers hope to develop an early diagnostic test for AD.

The study will include 170 participants between the ages of 60 and 80 years, some normal, some with MCI, some with mild AD, and some with frontotemporal dementia. After initial screening of volunteers, the researchers will give participants a complete baseline exam and 24-month follow-up exams over a period of five years.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, from all racial and ethnic categories between the ages of 60-80 years of age, with English as their first language.
* Residents of the New York City metropolitan area.
* Minimum of 12 years of education.
* Participants will be grouped according to the following classifications: normal aging, mild cognitive impairment (MCI), Alzheimer's disease (AD), or frontotemporal dementia (FTD).
* Participants will agree to ApoE genotyping and DNA banking.

Exclusion Criteria:

* Past history or MRI evidence of brain damage including significant trauma, stroke, hydrocephalus, lacunar infarcts, seizures, mental retardation or serious neurological disorder.
* Significant history of alcoholism or drug abuse.
* History of psychiatric illness (e.g., schizophrenia, mania or depression).
* Any focal signs or significant neuropathology.
* A score of 4 or greater on the Modified Hachinski Ischemia Scale suggesting cerebrovascular disease.
* A total score of 16 or more on the Hamilton Depression Scale to exclude possible cases of primary depression.
* Evidence of clinically relevant and uncontrolled hypertensive, cardiac, pulmonary, vascular, metabolic or hematologic conditions.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Hostility or refusal to cooperate.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that could be affected by the magnetic field employed during MRI imaging.
* History of familial early onset dementia.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2003-09; Study Completion 2008-08

CONTACTS AND LOCATIONS:
Overall Officials: Mony J. de Leon, Ed.D., Principal Investigator — Center for Brain Health, Silberstein Institute
Locations (1):
- Center for Brain Health, Silberstein Institute, New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] de Leon MJ, Segal S, Tarshish CY, DeSanti S, Zinkowski R, Mehta PD, Convit A, Caraos C, Rusinek H, Tsui W, Saint Louis LA, DeBernardis J, Kerkman D, Qadri F, Gary A, Lesbre P, Wisniewski T, Poirier J, Davies P. Longitudinal cerebrospinal fluid tau load increases in mild cognitive impairment. Neurosci Lett. 2002 Nov 29;333(3):183-6. doi: 10.1016/s0304-3940(02)01038-8. PMID 12429378
- [Background] Buerger K, Teipel SJ, Zinkowski R, Blennow K, Arai H, Engel R, Hofmann-Kiefer K, McCulloch C, Ptok U, Heun R, Andreasen N, DeBernardis J, Kerkman D, Moeller H, Davies P, Hampel H. CSF tau protein phosphorylated at threonine 231 correlates with cognitive decline in MCI subjects. Neurology. 2002 Aug 27;59(4):627-9. doi: 10.1212/wnl.59.4.627. PMID 12196665
- [Background] Mehta PD, Pirttila T, Mehta SP, Sersen EA, Aisen PS, Wisniewski HM. Plasma and cerebrospinal fluid levels of amyloid beta proteins 1-40 and 1-42 in Alzheimer disease. Arch Neurol. 2000 Jan;57(1):100-5. doi: 10.1001/archneur.57.1.100. PMID 10634455
- [Derived] Haghdel A, Smith N, Glodzik L, Li Y, Wang X, Crowder T, Zhu YS, Butler T, Blennow K, McIntire LB, Pahlajani S, Osborne J, Chiang G, de Leon M, Ivanidze J. Evidence of Pericyte Damage in a Cognitively Normal Cohort: Association With CSF and PET Biomarkers of Alzheimer Disease. Alzheimer Dis Assoc Disord. 2024 Apr-Jun 01;38(2):107-111. doi: 10.1097/WAD.0000000000000623. Epub 2024 May 16. PMID 38752577